CLINICAL TRIAL: NCT03381898
Title: Decreasing Health Disparities for Parkinson's Disease in Rural Communities: Assessing Feasibility of Coordinated Telehealth to Deliver Allied Health Care of Medication Management, Physical Therapy, and Speech Therapy
Brief Title: Telehealth Allied Health Care With People Who Have Parkinson's Disease Living in Rural Nevada and Wyoming
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wyoming (Other)
Collaborators: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1003674
Record Dates: First submitted 2017-11-29; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Parkinson Disease
Keywords: Telehealth; Physical therapy exercise; Speech therapy Lee Silverman voice treatment; Pharmacy medication management
MeSH Terms: conditions — Parkinson Disease | interventions — Speech Therapy

STUDY DESIGN:
Intervention Model Description: This is a feasibility and safety trial of a single arm a telehealth intervention (pharmacy, physical therapy, and speech therapy) to people with Parkinson's disease.
Masking Description: The outcomes assessment and the care providers will be blind to the aims of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth Coordinated Allied Health (Experimental): rural persons with Parkinson's disease will receive telehealth exercise, speech therapy, medication management for 8 weeks. Exercise, speech therapy, and medication management are usual care for persons with Parkinson's disease. Having the 3 areas coordinated in delivery via telehealth is the new delivery that our aims address
  Interventions: Behavioral: Telehealth Exercise, speech therapy, medication management

INTERVENTIONS:
Behavioral: Telehealth Exercise, speech therapy, medication management — Telehealth exercise once per week, speech therapy 4 times per week, medication management once per week

SUMMARY:
The investigators have developed a three-part allied health care intervention to be delivered via telehealth. These interventions are usually provided face-to-face. Telehealth access to healthcare is needed for people with Parkinson's disease living in rural locations, where providers are sparse and long travel times are often not feasible because of weather conditions, as well as the hallmark symptom of Parkinson's disease, movement disorders

DETAILED DESCRIPTION:
Parkinson's Disease & Allied Health. Parkinson's disease (PD), the second most common neurodegenerative disorder affecting more than a million people in the U.S., has no known cause or cure. Persons with PD use prescription medications and behavioral interventions to alleviate key problems such as walking, handling objects, and speaking. Individuals with PD, accessing multidisciplinary allied health care intervention, have shown functional gains. Without these ongoing, coordinated services, persons with PD become even more debilitated, and this can hasten a decline in their quality of life.

Parkinson's Disease & Rurality. For those in rural areas, there is a critical health disparity. People who live rurally contend with isolation. Wyoming and Nevada's population density are ranked 49th and 42nd. In conjunction with this low population density and mountainous terrain, individuals experience tremendous burdens including traveling long distances to see health care providers with expertise in treating PD. These factors contribute to the struggle of rural Americans with PD to manage this complicated, chronic disease.

Parkinson's Disease & Telehealth. Telehealth technology has successfully allowed the delivery of neurology care via "virtual house calls" with rural residents with PD. The virtual house call model was determined to be feasible and promising for specialist care in underserved rural areas. However, telehealth delivery of allied health care should also be examined.

Thus, the investigators propose an exploratory Phase 2 Behavioral Clinical Trial to determine feasibility, safety, and signal of efficacy for telehealth coordinated allied health care for persons with Parkinson's disease in rural Wyoming and Nevada. All 20 participants will be in one arm receiving telehealth exercise, speech therapy, and medication management for eight weeks.

Specific Aims:

For persons with Parkinson's disease in rural Wyoming and Nevada, the investigators will:

Aim 1 Test the feasibility of speech therapy, exercise therapy and medication management coordinated through telehealth.

Aim 2 Determine the safety of the coordinated telehealth speech therapy, exercise therapy, and medication management.

Aim 3 Measure signal of efficacy for telehealth outcomes

ELIGIBILITY:
Inclusion Criteria:

* Speak English
* Are 30 years or older
* Have been diagnosed with Parkinson's Disease by a primary care provider
* Allow for us to communicate about you to your primary care provider (i.e., physician, nurse practitioner, or physician assistant)
* Can stand alone for 10 min without holding on to anything
* Are taking at least one medication for Parkinson's Disease
* Are willing the participate in an 8-week study
* Will provide your physical address, your phone number, and an emergency contact's phone number for us to use if an emergency occurs during your telehealth session.

Exclusion Criteria:

* Have dementia or problems following directions
* Have a medical diagnosis that would limit exercises
* have experienced a fall that required physician evaluation (Emergency Department, urgent care or a hospitalization) within the past year
* Requires an assistive device or person (e.g., cane or walker) for walking, standing, balancing
* Currently use a structured exercise regimen defined as participation in a regular exercise program consisting of more than 60 minutes per week in total

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Feasibility of the 8-week telehealth program | 8 weeks
  The number of sessions completed and ability to use the necessary technology.
Aim 2: Safety of the 8-week telehealth program | 8 weeks
  The frequency and nature of adverse events during participation of the telehealth program.
Aim 3: Change in Signal of efficacy of the telehealth program - overall | 0, 8, 24 weeks
  The change in quality of life between baseline at the beginning of the study and after the 8 week intervention. In addition, change will also be measured between the end of the 8 week intervention and 18 weeks later (24 weeks from the baseline). This quality of life measures is a self-report, PD-specific Parkinson's Disease Questionnaire 39 (PDQ39). There are 39 items in 8 subsections (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, bodily discomfort). Each item ranges from 0 (never) to 4 (always). The overall score and subsection scores are calculated by taking the means of each item divided by the total for that section; thus, converting the score into a percentage with higher percentages equating to more disability.

SECONDARY OUTCOMES:
Aim 3: Signal of efficacy of the telehealth program - pharmacy | 8, 24 weeks
  Change in pill count (i.e., how many pills of each prescription are taken) over the period of the study.
Aim 3: Signal of efficacy of the telehealth program - physical therapy 1 | 0, 8, 24 weeks
  Change in 30 second Sit-to-Stand test which measures how many times the participant can stand in 30 seconds.
Aim 3: Signal of efficacy of the telehealth program - physical therapy 2 | 0, 8, 24 weeks
  Change in Parkinson's Fatigue Scale, which is a self-report measure of fatigue. This scale measures 16 items using a Likert scale with a low score of 16 (low fatigue) and a high score of 80 (high fatigue).
Aim 3: Signal of efficacy of the telehealth program - physical therapy 3 | 0, 8, 24 weeks
  Change in Unified Parkinson's Disease Rating Scale II (UPDRS II), which is a self-report of PD-specific motor aspects of experiences of daily living. There are 13 items with scores ranging from 0 (normal) to 4 (severe). Thus, a score of 0 indicates normal function whereas a score of 52 (the highest possible score) suggestive of severe motor deficits with activities of daily living.
Aim 3: Signal of efficacy of the telehealth program - speech therapy 1 | 0, 8, 24 weeks
  Change in self-report Communication Effectiveness Scale, which is an 8 question scale using a 4-point likert scale on how the participant social participation is affected by his speech and communication. The scores range from 0 (not effective) to 32 (very effective communication in all situations).
Aim 3: Signal of efficacy of the telehealth program - speech therapy 2 | 0, 8, 24 weeks
  Change in Vocal sound level intensity using the Lee Silverman Voice Treatment (LSVT) Companion Software which measures speech intensity. Changes in vocal sound level could range from - 6 decibel (dB) (reduced loudness) to at least + 6dB which is the average change and is perceptually noticeable.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jo Cooley Hidecker, PhD, Principal Investigator — University of Wyoming; Merrill Landers, DPT, Ph.D., Study Director — University of Nevada, Las Vegas
Locations (2):
- United States (2):
  - University of Nevada Las Vegas, Las Vegas, Nevada
  - University of Wyoming, Laramie, Wyoming

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study to help determine appropriate individual participant data (IPD) categories

REFERENCES:
- [Background] Ellis T, Katz DI, White DK, DePiero TJ, Hohler AD, Saint-Hilaire M. Effectiveness of an inpatient multidisciplinary rehabilitation program for people with Parkinson disease. Phys Ther. 2008 Jul;88(7):812-9. doi: 10.2522/ptj.20070265. Epub 2008 Apr 24. PMID 18436568
- [Background] Mather, M., Jacobsen, L.A., & Pollard, K.M. (2015). Aging in the United Sates. Population Bulletin 70
- [Background] Sapir S, Ramig L, Fox C. Speech and swallowing disorders in Parkinson disease. Curr Opin Otolaryngol Head Neck Surg. 2008 Jun;16(3):205-10. doi: 10.1097/MOO.0b013e3282febd3a. PMID 18475072
- [Background] Atkinson-Clement C, Sadat J, Pinto S. Behavioral treatments for speech in Parkinson's disease: meta-analyses and review of the literature. Neurodegener Dis Manag. 2015;5(3):233-48. doi: 10.2217/nmt.15.16. PMID 26107322
- [Background] Allen NE, Sherrington C, Suriyarachchi GD, Paul SS, Song J, Canning CG. Exercise and motor training in people with Parkinson's disease: a systematic review of participant characteristics, intervention delivery, retention rates, adherence, and adverse events in clinical trials. Parkinsons Dis. 2012;2012:854328. doi: 10.1155/2012/854328. Epub 2011 Nov 16. PMID 22191077
- [Background] Allen NE, Sherrington C, Paul SS, Canning CG. Balance and falls in Parkinson's disease: a meta-analysis of the effect of exercise and motor training. Mov Disord. 2011 Aug 1;26(9):1605-15. doi: 10.1002/mds.23790. Epub 2011 Jun 14. PMID 21674624
- [Background] Davis KL, Edin HM, Allen JK. Prevalence and cost of medication nonadherence in Parkinson's disease: evidence from administrative claims data. Mov Disord. 2010 Mar 15;25(4):474-80. doi: 10.1002/mds.22999. PMID 20131374
- [Background] Herd CP, Tomlinson CL, Deane KH, Brady MC, Smith CH, Sackley CM, Clarke CE. Comparison of speech and language therapy techniques for speech problems in Parkinson's disease. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD002814. doi: 10.1002/14651858.CD002814.pub2. PMID 22895931
- [Background] Miller N, Noble E, Jones D, Burn D. Life with communication changes in Parkinson's disease. Age Ageing. 2006 May;35(3):235-9. doi: 10.1093/ageing/afj053. Epub 2006 Mar 15. PMID 16540492
- [Background] Fox, C.M., & Ramig, L.O. (1997). Vocal sound pressure level and self-perception of speech and voice in men and women with idiopathic parkinson disease. Am J Speech Lang Pathol 6, 85-94
- [Background] Baumgartner CA, Sapir S, Ramig TO. Voice quality changes following phonatory-respiratory effort treatment (LSVT) versus respiratory effort treatment for individuals with Parkinson disease. J Voice. 2001 Mar;15(1):105-14. doi: 10.1016/s0892-1997(01)00010-8. PMID 12269625
- [Background] Ramig LO, Countryman S, O'Brien C, Hoehn M, Thompson L. Intensive speech treatment for patients with Parkinson's disease: short-and long-term comparison of two techniques. Neurology. 1996 Dec;47(6):1496-504. doi: 10.1212/wnl.47.6.1496. PMID 8960734
- [Background] Constantinescu G, Theodoros D, Russell T, Ward E, Wilson S, Wootton R. Treating disordered speech and voice in Parkinson's disease online: a randomized controlled non-inferiority trial. Int J Lang Commun Disord. 2011 Jan-Feb;46(1):1-16. doi: 10.3109/13682822.2010.484848. PMID 21281410
- [Background] Halpern AE, Ramig LO, Matos CE, Petska-Cable JA, Spielman JL, Pogoda JM, Gilley PM, Sapir S, Bennett JK, McFarland DH. Innovative technology for the assisted delivery of intensive voice treatment (LSVT(R)LOUD) for Parkinson disease. Am J Speech Lang Pathol. 2012 Nov;21(4):354-67. doi: 10.1044/1058-0360(2012/11-0125). Epub 2012 Oct 15. PMID 23071195
- [Background] Wight S, Miller N. Lee Silverman Voice Treatment for people with Parkinson's: audit of outcomes in a routine clinic. Int J Lang Commun Disord. 2015 Mar-Apr;50(2):215-25. doi: 10.1111/1460-6984.12132. Epub 2014 Dec 3. PMID 25469736
- [Background] Theodoros D, Russell TG, Hill A, Cahill L, Clark K. Assessment of motor speech disorders online: a pilot study. J Telemed Telecare. 2003;9 Suppl 2:S66-8. doi: 10.1258/135763303322596318. PMID 14728766
- [Background] Goodwin VA, Richards SH, Taylor RS, Taylor AH, Campbell JL. The effectiveness of exercise interventions for people with Parkinson's disease: a systematic review and meta-analysis. Mov Disord. 2008 Apr 15;23(5):631-40. doi: 10.1002/mds.21922. PMID 18181210
- [Background] Stempak, N. (2016). Physical therapy for Parkinson's: The balancing act of fall prevention involves cueing, exercise, and plenty of patience. Long-Term Living: For the Continuing Care Professional 65, 12.
- [Background] Geraedts H, Zijlstra A, Bulstra SK, Stevens M, Zijlstra W. Effects of remote feedback in home-based physical activity interventions for older adults: a systematic review. Patient Educ Couns. 2013 Apr;91(1):14-24. doi: 10.1016/j.pec.2012.10.018. Epub 2012 Nov 26. PMID 23194823
- [Background] Cipolle, R.J., Strand, L., and Morley, P.C. (2012). Pharmaceutical care practice: The patient-centered approach to medication management.(New York: McGraw-Hill)
- [Background] Shin JY, Habermann B. Medication Adherence in People With Parkinson Disease. J Neurosci Nurs. 2016 Jul-Aug;48(4):185-94. doi: 10.1097/JNN.0000000000000198. PMID 27224682
- [Background] Shin JY, Habermann B, Pretzer-Aboff I. Challenges and strategies of medication adherence in Parkinson's disease: A qualitative study. Geriatr Nurs. 2015 May-Jun;36(3):192-6. doi: 10.1016/j.gerinurse.2015.01.003. Epub 2015 Feb 26. PMID 25728485
- [Background] Ramalho de Oliveira D, Brummel AR, Miller DB. Medication therapy management: 10 years of experience in a large integrated health care system. J Manag Care Pharm. 2010 Apr;16(3):185-95. doi: 10.18553/jmcp.2010.16.3.185. PMID 20331323
- [Background] Ellis T, Boudreau JK, DeAngelis TR, Brown LE, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Dibble LE. Barriers to exercise in people with Parkinson disease. Phys Ther. 2013 May;93(5):628-36. doi: 10.2522/ptj.20120279. Epub 2013 Jan 3. PMID 23288910
- [Background] Dorsey ER, Vlaanderen FP, Engelen LJ, Kieburtz K, Zhu W, Biglan KM, Faber MJ, Bloem BR. Moving Parkinson care to the home. Mov Disord. 2016 Sep;31(9):1258-62. doi: 10.1002/mds.26744. Epub 2016 Aug 8. PMID 27501323
- [Background] Achey M, Aldred JL, Aljehani N, Bloem BR, Biglan KM, Chan P, Cubo E, Dorsey ER, Goetz CG, Guttman M, Hassan A, Khandhar SM, Mari Z, Spindler M, Tanner CM, van den Haak P, Walker R, Wilkinson JR; International Parkinson and Movement Disorder Society Telemedicine Task Force. The past, present, and future of telemedicine for Parkinson's disease. Mov Disord. 2014 Jun;29(7):871-83. doi: 10.1002/mds.25903. Epub 2014 May 17. PMID 24838316
- [Background] Hustad, K.C. (1999). Optimizing communicative effectiveness: Bringing it together. In Management of motor speech disorders in children and adults, K. Yorkston, D. Beukelman, E.A. Strand, andK.R. Bell, eds. (Austin, TX, Pro-Ed), pp 483-537
- [Background] Donovan NJ, Kendall DL, Young ME, Rosenbek JC. The communicative effectiveness survey: preliminary evidence of construct validity. Am J Speech Lang Pathol. 2008 Nov;17(4):335-47. doi: 10.1044/1058-0360(2008/07-0010). PMID 18957572
- [Background] Donovan, N.J., Velozo, C.A., Rosenbek, J.C. (2007). The communicative effectiveness survey: Investigating its item-level psychometrics. Journal of Medical Speech-Language Pathology 15, 433-447
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Brown RG, Dittner A, Findley L, Wessely SC. The Parkinson fatigue scale. Parkinsonism Relat Disord. 2005 Jan;11(1):49-55. doi: 10.1016/j.parkreldis.2004.07.007. PMID 15619463
- [Background] Gallagher DA, Lees AJ, Schrag A. Unified Parkinson's Disease Rating Scale (UPDRS) part I as a screening and diagnostic instrument for apathy in patients with Parkinson's disease. Parkinsonism Relat Disord. 2008 Nov;14(7):586-7. doi: 10.1016/j.parkreldis.2008.01.005. Epub 2008 Mar 6. No abstract available. PMID 18328769
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Haaxma CA, Bloem BR, Borm GF, Horstink MW. Comparison of a timed motor test battery to the Unified Parkinson's Disease Rating Scale-III in Parkinson's disease. Mov Disord. 2008 Sep 15;23(12):1707-17. doi: 10.1002/mds.22197. PMID 18649395
- [Background] McKinlay A, Grace RC, Dalrymple-Alford JC, Roger D, Anderson T, Fink J. The accuracy of the Unified Parkinson's Disease Rating Scale (UPDRS-Section 1) as a screening measure for depression. Parkinsonism Relat Disord. 2008;14(2):170-2. doi: 10.1016/j.parkreldis.2007.03.002. Epub 2007 May 4. No abstract available. PMID 17481937
- [Background] Pedersen KF, Larsen JP, Aarsland D. Validation of the Unified Parkinson's Disease Rating Scale (UPDRS) section I as a screening and diagnostic instrument for apathy in patients with Parkinson's disease. Parkinsonism Relat Disord. 2008;14(3):183-6. doi: 10.1016/j.parkreldis.2007.07.015. Epub 2007 Sep 21. PMID 17889589
- [Background] Stewart M. The validity of an interview to assess a patient's drug taking. Am J Prev Med. 1987 Mar-Apr;3(2):95-100. PMID 3330658
- [Background] Botelho RJ, Dudrak R 2nd. Home assessment of adherence to long-term medication in the elderly. J Fam Pract. 1992 Jul;35(1):61-5. PMID 1613477
- [Background] Choo PW, Rand CS, Inui TS, Lee ML, Cain E, Cordeiro-Breault M, Canning C, Platt R. Validation of patient reports, automated pharmacy records, and pill counts with electronic monitoring of adherence to antihypertensive therapy. Med Care. 1999 Sep;37(9):846-57. doi: 10.1097/00005650-199909000-00002. PMID 10493464
- [Background] Lee JK, Grace KA, Foster TG, Crawley MJ, Erowele GI, Sun HJ, Turner PT, Sullenberger LE, Taylor AJ. How should we measure medication adherence in clinical trials and practice? Ther Clin Risk Manag. 2007 Aug;3(4):685-90. PMID 18472991
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479